CLINICAL TRIAL: NCT07007234
Title: Sedentary Behavior and Depressive Symptoms: Influence of Specific Domains of Sedentary Behavior
Brief Title: Sedentary Behavior and Depressive Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Hamilton Augusto Roschel da Silva, PhD., University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 85919225.2.0000.0081
Record Dates: First submitted 2025-05-20; First posted 2025-06-05 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity intervention (Experimental): Patients allocated to this arm will be submitted to intervention (4-month goal-setting intervention aimed to replace mentally passive sedentary behaviors with mentally active sedentary behaviors, light physical activity, or moderate-to-vigorous activity)
  Interventions: Behavioral: Physical activity intervention
- Standard of care (Experimental): Patients allocated to this arm will be submitted to intervention (4 face-to-face individual sessions during 4 months, lasting ~15-30 minutes, however they will receive general instructions related to WHO guidelines for physical activity.)
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Physical activity intervention — The INTERVENTION group will participate in a 4-month goal-setting intervention aimed to replace mentally passive sedentary behaviors with mentally active sedentary behaviors, light physical activity, or moderate-to-vigorous activity.
  Arms: Physical activity intervention
Behavioral: Standard of care — The CONTROL group also will participate of 4 face-to-face individual sessions during the experimental period, lasting ~15-30 minutes, however they will receive general instructions related to WHO guidelines for physical activity
  Arms: Standard of care

SUMMARY:
Depressive symptoms are commonly observed in the general population. Individuals with subclinical forms of depression (e.g., not meet the criteria to major depression disorder) are at increased risk of mortality than the general population which is partially explained by the higher incidence of cardiovascular diseases. Currently, the effectiveness of the frontline treatment for depression is not consensual. Further, it also may be expensive for individuals with mild to moderate depression. Sedentary behavior is an independent risk factor for cardiometabolic diseases and mental disorders. However, recent evidence suggests that not all types of sedentary behavior are equally detrimental. For instance, mentally passive sedentary behavior (e.g., watching TV) appear to be detrimental for health outcomes whereas mentally active sedentary behavior (e.g., desk-based office work) appear to offer health benefits. However, more studies are required to determine the magnitude of association between distinct types of sedentary behaviors (e.g., watching TV, listening to music, talking while sitting, sitting around and doing nothing special) with depressive symptoms as well as randomized clinical trials investigating potential benefits of interventions to replace mentally-passive sedentary behaviors with mentally active sedentary behaviors, light physical activity or moderate-to-vigorous activity in individuals with mild to moderate depression. Therefore, the aim of this proposal is to investigate the influence of mentally passive sedentary behavior (i.e., watching TV, listening to music, talking while sitting, sitting around, and doing nothing special) on depressive symptoms. This is a randomized clinical trial. Participants with mild to severe depressive symptoms will be randomly assigned (1:1) into either INTERVENTION or CONTROL group, using a computer-generated randomization code. Depressive symptoms, quality of life, physical activity, sedentary behavior, body composition, and functionality will be assessed at baseline (PRE) and 4 (POST) months after the experimental period. The INTERVENTION group will participate in a 4-month goal-setting intervention aimed to replace mentally passive sedentary behaviors with mentally active sedentary behaviors, light physical activity, or moderate-to-vigorous activity while CONTROL group will receive general instructions related to WHO guidelines for physical activity.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged over 17 years;
* mild to severe depressive symptoms.

Exclusion Criteria:

* cancer in the past 5 years;
* inability to perform the physical tests;
* prior diagnosis of muscle degenerative disease (e.g., myopathies, amyotrophic lateral sclerosis);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms | Baseline (Pre-intervention) and 16 weeks (Post-intervention)
  The depressive symptoms will be assessed by Beck's Depressive Inventory (BDI). Score ranges from 0 to 63 points, being higher scores indicative of higher symptoms of depression.

SECONDARY OUTCOMES:
Anxiety Symptoms (primary outcome) | Baseline (Pre-intervention) and 16 weeks (Post-intervention)
  The anxiety symptoms will be assessed by Beck's Anxiety Inventory (BAI).Score ranges from 0 to 63 points, being higher scores indicative of higher symptoms of anxiety.
Indirect physical activity levels assessment | Baseline (Pre-intervention) and 16 weeks (Post-intervention)
  Indirect Physical activity levels will be assessed using the International Physical Activity Questionnaire-Long Form (IPAQ).
Objective physical activity levels assessment | Baseline (Pre-intervention) and 16 weeks (Post-intervention)
  Objective measures of physical activity levels will be assessed using ActiGraph GT9X® accelerometers
Indirect sedentary behavior assessment | Baseline (Pre-intervention) and 16 weeks (Post-intervention)
  Indirect levels of sedentary behavior will be assessed using the questionnaire LASA-SBQ (i.e., Longitudinal Aging Study Amsterdam - Sedentary Behavior Questionnaire).
Objective sedentary behavior assessment | Baseline (Pre-intervention) and 16 weeks (Post-intervention)
  The objective measures of sedentary time will be assessed using ActiGraph GT9X® accelerometers.
Quality of life assessement | Baseline (Pre-intervention) and 16 weeks (Post-intervention)
  The quality of life will be assessed using the WHOQOL-bref. Score ranges from 0 to 100 points, being higher scores indicative of higher quality of life.
Body Weight | Baseline (Pre-intervention) and 16 weeks (Post-intervention)
  Body weight will be assessed on a calibrated digital scale.
Fat mass (kg) | Baseline (Pre-intervention) and 16 weeks (Post-intervention)
  Fat mass (kg) will be assessed using 4-point bioelectrical impedance device (hands and feet).
Fat-free mass (kg) | Baseline (Pre-intervention) and 16 weeks (Post-intervention)
  Fat-free mass (kg) will be assessed using 4-point bioelectrical impedance device (hands and feet).
Muscle Function (30-s Sit-to-stand Test) | Baseline (Pre-intervention) and 16 weeks (Post-intervention)
  The 30-second sit-to-stand test is a simple measure of lower body strength and functional capacity. Participants are asked to rise from a seated position and sit back down as many times as possible within 30 seconds. The total number of complete sit-to-stand repetitions performed in the given time is recorded. This test is commonly used to assess physical fitness and mobility, particularly in older adults or individuals with health conditions.
Muscle Function (Timed-up-and-go) | Baseline (Pre-intervention) and 16 weeks (Post-intervention)
  The Timed Up and Go (TUG) test is a simple and widely used assessment of mobility and balance. Participants are asked to stand up from a seated position, walk 3 meters, turn around, walk back to the chair, and sit down again, all as quickly as possible. The total time taken to complete the task is recorded. The TUG test is commonly used to evaluate functional mobility, fall risk, and the ability to perform daily activities, particularly in older adults or individuals with mobility impairments.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - University of Santo Amaro, São Paulo, SO
  - University Santo Amaro, São Paulo, São Paulo